CLINICAL TRIAL: NCT03015077
Title: Impacts of Oral Supplement With L-Glutamine on the Radiation-induced Toxicity and Nutritional Status of Head and Neck Cancer Patients Under Radiotherapy
Brief Title: Effects of Oral L-Glutamine in Head and Neck Cancer Patients During Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: KMUHIRB-2014-12-01(II)
Record Dates: First submitted 2016-12-11; First posted 2017-01-09 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2015-02

CONDITIONS: Head and Neck Cancer
Keywords: Glutamine
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Glutamine; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glutamine (Active Comparator): intake of 5g glutamine and 10g maltodextrin. Oral glutamine is a food additive issued by food and drug government in Taiwan with number 009929.L-Glutamine and maltodextrin are both nutritional supplements. In the glutamine arm: 10 g L-Glutamine and 5 g maltodextrin.
  The patients take their supplements three times a day during the period: 7 days before radiotherapy to 14 days after radiotherapy.
  Interventions: Dietary Supplement: oral glutamine; Radiation: Radiotherapy
- placebo (Placebo Comparator): intake of 15g maltodextrin. The patients take their supplements three times a day during the period: 7 days before radiotherapy to 14 days after radiotherapy.
  Interventions: Dietary Supplement: placebo; Radiation: Radiotherapy

INTERVENTIONS:
Dietary Supplement: oral glutamine — L-Glutamine and maltodextrin are both nutritional supplements. In the glutamine arm: 10 g L-Glutamine and 5 g maltodextrin. The patients take their supplements three times a day during the period: 7 days before radiotherapy to 14 days after radiotherapy.
  Arms: Glutamine
Dietary Supplement: placebo — in the placebo arm: 15 g maltodextrin. The patients take their supplements three times a day during the period: 7 days before radiotherapy to 14 days after radiotherapy.
  Arms: placebo
Radiation: Radiotherapy — All patients undergo radiotherapy. 5 days a week. All patients had a dental evaluation for good oral hygiene prior to computed tomography simulation for radiotherapy. Post-operative patients received planned course of adjuvant treatment of 60 to 66 Gy in 2-Gy fractions to the surgical bed. The course of radiation was initiated no more than 6 weeks after resection. Patients without operation received definitive treatment to 70 Gy in 2-Gy fractions.

SUMMARY:
The rapidly increasing mortality and incidence of oral cancer has become a public health major problem in Taiwan. To date, the treatment of head and neck cancer mainly include surgery, radiotherapy and chemotherapy. However, radiotherapy and chemotherapy might have an influence on the patients' diet by causing dismal side effects, including nausea, vomiting, pain, infection, dysorexia, allotriogeustia, oral ulceration and dysphagia, which make the patients more difficult to absorb nutrients. In the previous study, the incidence of malnutrition among the patients with cancer has been estimated at between 40 and 80%, especially occurred in the patients with head and neck cancers and upper gastrointestinal cancers.

In this study, the effect of supplement with L-Glutamine on the nutritional status and radiation-induced toxicity of head and neck cancer patients will be evaluated to improve the patients' quality of life when they are undergoing radiotherapy. When the head and neck cancer patients undergoing radiotherapy, patients' instructions and nutrient intervention of L-Glutamine are performed to maintain the patients' nutritional status and reduce the patients' diet-related or other side effects caused by radiotherapy. It is anticipated that head and neck cancer patients with surgery and radiotherapy intake with L-Glutamine might decrease treatment-related side effects and hence improve their quality of life when they are undergoing radiotherapy.

DETAILED DESCRIPTION:
1. Written informed consent must be obtained before any study specific procedures are undertaken.
2. The process of the experiment A. head and neck cancer patients with surgery and radiotherapy are identified in clinic at the Department of Dentistry and the Department of Radiotherapy in Kaohsiung Medical University Chung-Ho Memorial Hospital.

B. Inform these patients about the value of this clinical trial in detail, and make sure that they understand all the meanings of each procedure in this clinical trial. Subsequently, the patients who are willing to participate in this study are enrolled after completing institutionally approved informed consent.

C. In order to assess the effect of supplement with L-Glutamine on the nutritional status and diet of head and neck cancer patients with surgery and radiotherapy, the enrolled patients will be divided into two groups randomly. One group is supplied with 10 g L-Glutamine and 5 g maltodextrin; the other group is supplied with 15 g maltodextrin as control group. The patients of these two groups take their supplemental nutrients three times a day, respectively, in a period of time of 7 days before radiotherapy to 14 days after radiotherapy.

D. Meanwhile, the research assistants will monitor the patients' condition carefully by recording their daily diet, nutritional status and side effects caused by radiotherapy at three specific time-points during the whole clinic trial program course.

E. The monitor items of patients' nutritional status include the daily diet of patients before and after radiotherapy by recording 24 hr recall table and food frequency table,(b) the physical examination of height, weight, ideal weight, tricept skinfold (TSF), mid-arm circumference (MAC) and mid-arm muscle circumference (MAMC), (d) prognostic nutritional index (PNI), (e) biochemistry inspection assessment and (g) complete blood count (CBC).

F. The monitor items of patients' diet-related side effects caused by radiotherapy include (a) oral mucositis and (b) neck dermatitis.

G. The above-mentioned monitor items will be recorded carefully by the research assistants at three specific time-points during the whole clinic trial program course, which are initial point (7 days before radiotherapy), medium point (medium date during radiotherapy) and final point (14 days after radiotherapy).

H. The research assistants will help the patients make an appointment, and let them visit the doctor on schedule. And make sure the patients actually follow up the suggestions and obey the instructions during the clinic trial.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological diagnosis of malignant head and neck tumor.
* able to open his or her mouth wider than the width of one finger during the assessment of oral mucositis.
* Eastern Cooperative Oncology Group（ECOG）0-2
* complete radiotherapy (six to seven weeks with targets involving oral cavity or oropharynx)

Exclusion Criteria:

* History of previous radiotherapy.
* diabetes or nephritic or hepatic problems.
* serious infection or sepsis.
* distant metastases

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
grade of oral mucositis | once a week during radiotherapy and once after radiotherapy up to 8 weeks
  Oral mucositis and radiation-induced dermatological toxicity were evaluated during and after treatment using the National Cancer Institute Common Toxicity Criteria version 3.0 (CTCAE v.3). The scoring was done as the patients went through the treatment by the attending physicians. Post-operative patients received planned course of adjuvant treatment of 60 to 66 Gy in 2-Gy fractions to the surgical bed. Patients without operation received definitive treatment to 70 Gy in 2-Gy fractions.
grade of neck dermatitis | once a week during radiotherapy and once after radiotherapy up to 8 weeks
  Oral mucositis and radiation-induced dermatological toxicity were evaluated during and after treatment using the National Cancer Institute Common Toxicity Criteria version 3.0 (CTCAE v.3). The scoring was done as the patients went through the treatment by the attending physicians. Post-operative patients received planned course of adjuvant treatment of 60 to 66 Gy in 2-Gy fractions to the surgical bed. Patients without operation received definitive treatment to 70 Gy in 2-Gy fractions.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsihung Medical University Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Ottery FD. Cancer cachexia: prevention, early diagnosis, and management. Cancer Pract. 1994 Mar-Apr;2(2):123-31. PMID 8055014
- [Result] Adelstein DJ, Saxton JP, Lavertu P, Rybicki LA, Esclamado RM, Wood BG, Strome M, Carroll MA. Maximizing local control and organ preservation in stage IV squamous cell head and neck cancer With hyperfractionated radiation and concurrent chemotherapy. J Clin Oncol. 2002 Mar 1;20(5):1405-10. doi: 10.1200/JCO.2002.20.5.1405. PMID 11870186
- [Result] Bauer J, Capra S, Ferguson M. Use of the scored Patient-Generated Subjective Global Assessment (PG-SGA) as a nutrition assessment tool in patients with cancer. Eur J Clin Nutr. 2002 Aug;56(8):779-85. doi: 10.1038/sj.ejcn.1601412. PMID 12122555
- [Result] Cooper JS, Pajak TF, Forastiere AA, Jacobs J, Campbell BH, Saxman SB, Kish JA, Kim HE, Cmelak AJ, Rotman M, Machtay M, Ensley JF, Chao KS, Schultz CJ, Lee N, Fu KK; Radiation Therapy Oncology Group 9501/Intergroup. Postoperative concurrent radiotherapy and chemotherapy for high-risk squamous-cell carcinoma of the head and neck. N Engl J Med. 2004 May 6;350(19):1937-44. doi: 10.1056/NEJMoa032646. PMID 15128893
- [Result] Duncan M, Grant G. Oral and intestinal mucositis - causes and possible treatments. Aliment Pharmacol Ther. 2003 Nov 1;18(9):853-74. doi: 10.1046/j.1365-2036.2003.01784.x. PMID 14616150
- [Result] Forastiere A, Koch W, Trotti A, Sidransky D. Head and neck cancer. N Engl J Med. 2001 Dec 27;345(26):1890-900. doi: 10.1056/NEJMra001375. No abstract available. PMID 11756581
- [Result] Fukui T, Itoh Y, Orihara M, Yoshizawa K, Takeda H, Kawada S, Yoshioka T. [Elental prevented and reduced oral mucositis during chemotherapy in patients esophageal cancer]. Gan To Kagaku Ryoho. 2011 Dec;38(13):2597-601. Japanese. PMID 22189225
- [Result] Ogata Y, Takeuchi M, Ishibashi N, Kibe S, Takahashi K, Uchida S, Murakami N, Yahara T, Shirouzu K. [Efficacy of Elental on prevention for chemotherapy-induced oral mucositis in colorectal cancer patients]. Gan To Kagaku Ryoho. 2012 Apr;39(4):583-7. Japanese. PMID 22504682
- [Result] Ottery FD. Definition of standardized nutritional assessment and interventional pathways in oncology. Nutrition. 1996 Jan;12(1 Suppl):S15-9. doi: 10.1016/0899-9007(96)90011-8. PMID 8850213
- [Result] Paccagnella A, Morello M, Da Mosto MC, Baruffi C, Marcon ML, Gava A, Baggio V, Lamon S, Babare R, Rosti G, Giometto M, Boscolo-Rizzo P, Kiwanuka E, Tessarin M, Caregaro L, Marchiori C. Early nutritional intervention improves treatment tolerance and outcomes in head and neck cancer patients undergoing concurrent chemoradiotherapy. Support Care Cancer. 2010 Jul;18(7):837-45. doi: 10.1007/s00520-009-0717-0. Epub 2009 Aug 30. PMID 19727846
- [Result] Ravasco P, Monteiro Grillo I, Camilo M. Cancer wasting and quality of life react to early individualized nutritional counselling! Clin Nutr. 2007 Feb;26(1):7-15. doi: 10.1016/j.clnu.2006.10.005. Epub 2006 Dec 12. PMID 17166637
- [Result] Vidal-Casariego A, Calleja-Fernandez A, Ballesteros-Pomar MD, Cano-Rodriguez I. Efficacy of glutamine in the prevention of oral mucositis and acute radiation-induced esophagitis: a retrospective study. Nutr Cancer. 2013;65(3):424-9. doi: 10.1080/01635581.2013.765017. PMID 23530642
- [Result] Savarese DM, Savy G, Vahdat L, Wischmeyer PE, Corey B. Prevention of chemotherapy and radiation toxicity with glutamine. Cancer Treat Rev. 2003 Dec;29(6):501-13. doi: 10.1016/s0305-7372(03)00133-6. PMID 14585260
- [Result] van Bokhorst-de van der Schuer, van Leeuwen PA, Kuik DJ, Klop WM, Sauerwein HP, Snow GB, Quak JJ. The impact of nutritional status on the prognoses of patients with advanced head and neck cancer. Cancer. 1999 Aug 1;86(3):519-27. PMID 10430262
- [Result] Westin T, Jansson A, Zenckert C, Hallstrom T, Edstrom S. Mental depression is associated with malnutrition in patients with head and neck cancer. Arch Otolaryngol Head Neck Surg. 1988 Dec;114(12):1449-53. doi: 10.1001/archotol.1988.01860240099032. PMID 3190874
- [Result] Lacey JM, Wilmore DW. Is glutamine a conditionally essential amino acid? Nutr Rev. 1990 Aug;48(8):297-309. doi: 10.1111/j.1753-4887.1990.tb02967.x. PMID 2080048
- [Result] Buchman AL. Glutamine: is it a conditionally required nutrient for the human gastrointestinal system? J Am Coll Nutr. 1996 Jun;15(3):199-205. doi: 10.1080/07315724.1996.10718590. PMID 8935435
- [Result] Gibson RJ, Keefe DM, Lalla RV, Bateman E, Blijlevens N, Fijlstra M, King EE, Stringer AM, van der Velden WJ, Yazbeck R, Elad S, Bowen JM; Mucositis Study Group of the Multinational Association of Supportive Care in Cancer/International Society of Oral Oncology (MASCC/ISOO). Systematic review of agents for the management of gastrointestinal mucositis in cancer patients. Support Care Cancer. 2013 Jan;21(1):313-26. doi: 10.1007/s00520-012-1644-z. Epub 2012 Nov 10. PMID 23142924
- [Result] Kucuktulu E, Guner A, Kahraman I, Topbas M, Kucuktulu U. The protective effects of glutamine on radiation-induced diarrhea. Support Care Cancer. 2013 Apr;21(4):1071-5. doi: 10.1007/s00520-012-1627-0. Epub 2012 Oct 14. PMID 23064902
- [Result] Choi K, Lee SS, Oh SJ, Lim SY, Lim SY, Jeon WK, Oh TY, Kim JW. The effect of oral glutamine on 5-fluorouracil/leucovorin-induced mucositis/stomatitis assessed by intestinal permeability test. Clin Nutr. 2007 Feb;26(1):57-62. doi: 10.1016/j.clnu.2006.07.003. Epub 2006 Sep 1. PMID 16949180
- [Result] Stokman MA, Spijkervet FK, Boezen HM, Schouten JP, Roodenburg JL, de Vries EG. Preventive intervention possibilities in radiotherapy- and chemotherapy-induced oral mucositis: results of meta-analyses. J Dent Res. 2006 Aug;85(8):690-700. doi: 10.1177/154405910608500802. PMID 16861284
- [Result] Savarese D, Al-Zoubi A, Boucher J. Glutamine for irinotecan diarrhea. J Clin Oncol. 2000 Jan;18(2):450-1. doi: 10.1200/JCO.2000.18.2.450. No abstract available. PMID 10637264
- [Result] Kozelsky TF, Meyers GE, Sloan JA, Shanahan TG, Dick SJ, Moore RL, Engeler GP, Frank AR, McKone TK, Urias RE, Pilepich MV, Novotny PJ, Martenson JA; North Central Cancer Treatment Group. Phase III double-blind study of glutamine versus placebo for the prevention of acute diarrhea in patients receiving pelvic radiation therapy. J Clin Oncol. 2003 May 1;21(9):1669-74. doi: 10.1200/JCO.2003.05.060. PMID 12721240
- [Result] Ziegler TR, Benfell K, Smith RJ, Young LS, Brown E, Ferrari-Baliviera E, Lowe DK, Wilmore DW. Safety and metabolic effects of L-glutamine administration in humans. JPEN J Parenter Enteral Nutr. 1990 Jul-Aug;14(4 Suppl):137S-146S. doi: 10.1177/0148607190014004201. PMID 2119459
- [Result] Mahdavi R, Faramarzi E, Mohammad-Zadeh M, Ghaeammaghami J, Jabbari MV. Consequences of radiotherapy on nutritional status, dietary intake, serum zinc and copper levels in patients with gastrointestinal tract and head and neck cancer. Saudi Med J. 2007 Mar;28(3):435-40. PMID 17334475
- [Result] Kuhn KS, Muscaritoli M, Wischmeyer P, Stehle P. Glutamine as indispensable nutrient in oncology: experimental and clinical evidence. Eur J Nutr. 2010 Jun;49(4):197-210. doi: 10.1007/s00394-009-0082-2. Epub 2009 Nov 21. PMID 19936817
- [Result] Cockerham MB, Weinberger BB, Lerchie SB. Oral glutamine for the prevention of oral mucositis associated with high-dose paclitaxel and melphalan for autologous bone marrow transplantation. Ann Pharmacother. 2000 Mar;34(3):300-3. doi: 10.1345/aph.19168. PMID 10917373
- [Result] Muscaritoli M, Micozzi A, Conversano L, Martino P, Petti MC, Cartoni C, Cascino A, Rossi-Fanelli F. Oral glutamine in the prevention of chemotherapy-induced gastrointestinal toxicity. Eur J Cancer. 1997 Feb;33(2):319-20. doi: 10.1016/s0959-8049(96)00419-4. No abstract available. PMID 9135511
- [Result] Sharma R, Tobin P, Clarke SJ. Management of chemotherapy-induced nausea, vomiting, oral mucositis, and diarrhoea. Lancet Oncol. 2005 Feb;6(2):93-102. doi: 10.1016/S1470-2045(05)01735-3. PMID 15683818
- [Result] Diestel CF, Marques RG, Lopes-Paulo F, Paiva D, Horst NL, Caetano CE, Portela MC. Role of L-glutamine and glycine supplementation on irradiated colonic wall. Int J Colorectal Dis. 2007 Dec;22(12):1523-9. doi: 10.1007/s00384-007-0341-8. Epub 2007 Aug 10. PMID 17690894
- [Result] Xue H, Sawyer MB, Field CJ, Dieleman LA, Baracos VE. Nutritional modulation of antitumor efficacy and diarrhea toxicity related to irinotecan chemotherapy in rats bearing the ward colon tumor. Clin Cancer Res. 2007 Dec 1;13(23):7146-54. doi: 10.1158/1078-0432.CCR-07-0823. PMID 18056195
- [Result] Chattopadhyay S, Saha A, Azam M, Mukherjee A, Sur PK. Role of oral glutamine in alleviation and prevention of radiation-induced oral mucositis: A prospective randomized study. South Asian J Cancer. 2014 Jan;3(1):8-12. doi: 10.4103/2278-330X.126501. PMID 24665438
- [Derived] Huang CJ, Huang MY, Fang PT, Chen F, Wang YT, Chen CH, Yuan SS, Huang CM, Luo KH, Chuang HY, Wang YY, Lee HH. Randomized double-blind, placebo-controlled trial evaluating oral glutamine on radiation-induced oral mucositis and dermatitis in head and neck cancer patients. Am J Clin Nutr. 2019 Mar 1;109(3):606-614. doi: 10.1093/ajcn/nqy329. PMID 30753262